CLINICAL TRIAL: NCT03661671
Title: Application of Linked Color Imaging（LCI） in Diagnosis of Early Gastric Cancer(EGC): a Multicenter,Prospective, Randomized Controlled Study
Brief Title: Application of Linked Color Imaging（LCI） in Diagnosis of Early Gastric Cancer(EGC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanxi Province Cancer Hospital (Other); First People's Hospital of Hangzhou (Other); 307 Hospital of PLA (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Zhongshan Hospital Xiamen University (Other); Chongqing University Cancer Hospital (Other); Guilin Medical University, China (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Xiangya Hospital of Central South University (Other); Wuhan University (Other); Xi'an Central Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LCI2018
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Early Gastric Cancer
Keywords: Linked-color imaging; Detection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCI+white light (Experimental): Using white light firstly to observe from cardia to duodenum and then switch LCI model to observe from antrum to cardia
  Interventions: Diagnostic Test: LCI+white light
- White light (No Intervention): Using white light only.

INTERVENTIONS:
Diagnostic Test: LCI+white light — Firstly use white light to observe from cardia to duodenum and then switch LCI model to observe from antrum to cardia
  Arms: LCI+white light

SUMMARY:
the purpose of this study is to evaluate application value of LCI in the diagnosis of early gastric cancer.

DETAILED DESCRIPTION:
The detection rate of early gastric cancer is still very low in China. The investigators need a new and effective screening method to improve the detection rate. LCI (linked-color imaging)is a new model of laser endoscopy which can provide brighter image. LCI can provide clear image which can make red part redder and white part whiter, so suspicious lesion could be found easier. The study of this randomized controlled trial is to discuss effectiveness of LCI in the diagnosis of early gastric cancer and to find a new method to improve the detection rate of early gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk group of gastric cancer: H. pylori infection; previously suffering from chronic atrophic gastritis, intestinal metaplasia, gastric ulcer, gastric polyps, residual stomach after surgery, hypertrophic gastritis, malignant anemia and other precancerous diseases of gastric cancer;
2. First degree relatives of patients with gastric cancer;
3. There are other high risk factors for gastric cancer (high salt, salted diet, smoking, heavy drinking, etc.).
4. Patients with early gastric cancer treated with endoscopic therapy (ESD, EMR).
5. The informed consent has been signed.

Exclusion Criteria:

1. The TNM classification of cancer is consistent with those diagnosed by T2 above.
2. Patients with abnormal blood coagulation function or taking anticoagulants can not biopsy.
3. There were contraindications for gastroscopy.
4. A patient without self judgement;
5. Those who did not sign informed consent.
6. Previous gastroscopy has found suspicious lesions requiring careful examination.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of gastric neoplastic lesion | immediately following the procedure
  Include early gastric caner,high grade dysplasia low grade dysplasia and adenoma

SECONDARY OUTCOMES:
Specificity of detecting gastric neoplastic lesion | immediately following the procedure
  Include early gastric caner,high grade dysplasia low grade dysplasia and adenoma
Sensitivity of detecting gastric neoplastic lesion | immediately following the procedure
  Include early gastric caner,high grade dysplasia low grade dysplasia and adenoma

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Second Military Medical University
Locations (1):
- Department of Gastroenterology, Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fukuda H, Miura Y, Hayashi Y, Takezawa T, Ino Y, Okada M, Osawa H, Lefor AK, Yamamoto H. Linked color imaging technology facilitates early detection of flat gastric cancers. Clin J Gastroenterol. 2015 Dec;8(6):385-9. doi: 10.1007/s12328-015-0612-9. Epub 2015 Nov 11. PMID 26560036
- [Result] Okada M, Sakamoto H, Takezawa T, Hayashi Y, Sunada K, Lefor AK, Yamamoto H. Laterally Spreading Tumor of the Rectum Delineated with Linked Color Imaging Technology. Clin Endosc. 2016 Mar;49(2):207-8. doi: 10.5946/ce.2015.077. Epub 2016 Feb 12. No abstract available. PMID 26867550
- [Result] Sun X, Dong T, Bi Y, Min M, Shen W, Xu Y, Liu Y. Linked color imaging application for improving the endoscopic diagnosis accuracy: a pilot study. Sci Rep. 2016 Sep 19;6:33473. doi: 10.1038/srep33473. PMID 27641243